CLINICAL TRIAL: NCT00308490
Title: Phase IV Study of Iron Indices' Kinetics in Hemodialysis Patients
Brief Title: Changes in Iron Markers Following Iron Loading in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Papageorgiou General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 48/31-1-2005
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2006-09

CONDITIONS: Anemia in Chronic Renal Disease
MeSH Terms: interventions — Ferric Oxide, Saccharated

INTERVENTIONS:
Drug: iron sucrose

SUMMARY:
The purpose of this study is to describe alterations of serum ferritin, transferrin saturation, soluble transferrin receptor, % hypochromic erythrocytes, % reticulocytes, reticulocyte hemoglobin content after iron loading in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis for three months minimum
* stable epoetin dose for two months minimum
* serum ferritin concentration < 1000 ng/ml
* transferrin saturation < 50%
* parathormone concentration < 800 pg/ml

Exclusion Criteria:

* hemoglobin concentration > 13g/dl
* serum ferritin concentration < 20 ng/ml
* vitamin B12 and/or folic deficiency
* other hematologic disease than anemia
* cancer
* hypothyroidism
* infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-09; Study Completion 2007-01

PRIMARY OUTCOMES:
Ferritin alterations after iron loading at six and twelve weeks from the beginning of iron loading.

SECONDARY OUTCOMES:
All iron indices' alterations during twelve weeks from the beginning of iron loading.

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Mitsopoulos, MD, Principal Investigator — Papageorgiou General Hospital
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece